CLINICAL TRIAL: NCT02084121
Title: Allogeneic Stem Cell Transplantation for the Treatment of Multiple Sclerosis (Compassionate Use)
Status: No longer available | Type: Expanded Access
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: ICT-13080-Compassionate Use
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Metachromatic Leukodystrophy
Keywords: metachromatic leukodystrophy
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Enriched Hematopoetic Stem Cell Infusion — Enriched Hematopoetic Stem Cell Infusion

SUMMARY:
A subject was treated under compassionate use provisions under this study with facilitating cell therapy (FCRx) product manufactured using the CliniMACS (Miltenyi Biotec) device, rather than the Max Sep (Baxter) device.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of inherited metabolic disorder / inborn error of metabolism. Diagnosis should be confirmed by appropriate test(s) (enzyme and/or mutation analysis) before study entry. Patients must not be eligible for myeloablative chemotherapy as a preparative regimen for transplant due to age, co-morbidities or organ dysfunction.

   Inborn errors of metabolism / Inherited Metabolic Disorders (IMD) eligible for this Compassionate Use Provision include Metachromatic Leukodystrophy (MLD)
2. Patients must be ≥ 3 years of age
3. Patients must have Lansky or Karnofsky performance status ≥40
4. Patients must have adequate function of other organ systems as measured by:

   * Creatinine < 2.0 mg/dl and creatinine clearance ≥60 cc/min/1.73m2. Newborns must have a creatinine clearance > 25 cc/min. For babies < 3 months of age, the raw value on glomerular filtration rate (GFR) must be > 1 cc/kg/min.
   * Hepatic transaminases (ALT/AST) ≤4 x normal, bilirubin <2.0mg/dl
   * Normal cardiac function by echocardiogram or radionuclide scan (ejection fraction or shortening fraction >80% of normal value for age)
   * Pulmonary function tests demonstrating forced expiratory volume at one second (FEV1) of >50% of predicted for age. If child is too young for pulmonary function tests (PFTs), crying vital capacity result of >50% of normal value for age or resting pulse oximeter >85% on room air or clearance by pulmonologist will be required.
5. Patient must have a related donor [identical or mismatched for 1, 2 or 3 histocompatibility leukocyte antigen (HLA)-A, -B or -DR loci].
6. Patient, and parent, or legal guardian must have given written informed consent according to FDA guidelines.
7. Patients must have a minimum life expectancy of at least 6 months.
8. Female patients of childbearing potential cannot be pregnant or lactating/breast-feeding and must be either surgically sterile, postmenopausal (no menses for the previous 12 months), or must be practicing an effective method of birth control as determined by the investigator (e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy).

Exclusion Criteria:

* Patients with uncontrolled seizures, apnea, evidence of recurrent or uncontrolled aspiration, or need for chronic mechanical ventilation.
* Patients with allogeneic stem cell transplant with cytoreductive therapy in the past 6 months.
* Subjects must not have had previous radiation therapy that would preclude total body irradiation (TBI) (as determined by radiation therapist)
* Uncontrolled infection or severe concomitant diseases, which in the judgment of the Principal Investigator, could not tolerate reduced intensity transplantation.
* Severe impairment of functional performance as evidenced by a Karnofsky (patients >16 years old) or Lansky (children <16 years old) score <40%
* Subjects with a positive human immunodeficiency virus (HIV) antibody test result
* Subjects who are pregnant, as indicated by a positive serum human chorionic gonadotropin (HCG) test
* Subjects whose only donor is pregnant at the time of intended transplant
* Subjects of childbearing potential who are not practicing adequate contraception as defined by the investigator at the site
* Jehovah's witness
* Patients that have any comorbid condition which, in the view of the Principal Investigators, renders the patient at too high a risk from treatment complications and regimen related morbidity/mortality.
* Lack of related donors

Min Age: 3 Years | Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States